CLINICAL TRIAL: NCT04715698
Title: Effectiveness of A Hemodynamic-Guided Treatment Strategy to Improve Blood Pressure Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Collaborators: Yale University (Other); Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Ningling Sun, Director of Hypertension Department at Heart Center, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20181201
Record Dates: First submitted 2021-01-11; First posted 2021-01-20 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Hypertension
Keywords: Hypertension; ICG-guided; Hemodynamic profiling; Impedance cardiography
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ICG-guided (Experimental): anti-hypertensive drug selection based on physician's experience and hemodynamic profiling by measured ICG
  Interventions: Other: ICG-guided drug selection
- Empirical (Active Comparator): anti-hypertensive drug selection based on physician's experience only
  Interventions: Other: empirical drug selection

INTERVENTIONS:
Other: ICG-guided drug selection — anti-hypertensive drug selection based on patient's hemodynamic profiling and physician's experience
  Arms: ICG-guided
Other: empirical drug selection — anti-hypertensive drug selection based on physician's experience only
  Arms: Empirical

SUMMARY:
A single-center, single-blind, randomized study to investigate the effectiveness of a hemodynamic-guided treatment strategy to improve blood pressure control

DETAILED DESCRIPTION:
Hypertension is a hemodynamic-related disorder characterized by abnormalities of the cardiac output (CO) and/or systemic vascular resistance (SVR). It is hypothesized that selecting antihypertensive therapy based on patients' hemodynamic profile could lead to more effective blood pressure (BP) control than standard care in a real-world population of hypertensive patients in outpatient setting. A single-center, randomized trial was conducted to include adults with uncontrolled hypertension who seek outpatient care at Peking University People's Hospital between December 2018 and December 2019 in Beijing, China.

Participants were randomly assigned to the standard care group or the hemodynamic group in a 1:1 ratio. Impedance cardiography (ICG) was performed with all participants to measure hemodynamic parameters. Only physicians in the hemodynamic group were provided with patients' ICG findings and a computerized clinical decision support of recommended treatment choices based on patients' hemodynamic profiles. The primary outcomes were the reductions in systolic BP (SBP) and diastolic BP (DBP) levels at the follow-up visit 8(±4) weeks after baseline. Secondary outcomes included achievement of BP goal of <140/ 90 mmHg and the reductions in BP by baseline BP, age, sex, and BMI.

The ICG device used (HDproTM CHM T3002/P3005, designed by Beijing Li-Heng Medical Technologies, Ltd, manufactured by Shandong Baolihao Medical Appliances, Ltd.) was developed based on improved hardware and advanced digital filtering algorithms, and has been validated versus both invasive thermodilution and non-invasive echocardiography in different settings.

ELIGIBILITY:
Inclusion Criteria:

1. office BP >= 140/90 mmHg
2. hypertensive patients who were treatment naive or previously treated with 1-3 anti-hypertensives
3. age 18-85, males or females
4. agree to sign informed consent

Exclusion Criteria:

1. having unstable hemodynamics diseases, or had myocardial infarction (MI), heart failure (HF) or chronic kidney disease (CKD) within previous 6 months
2. using large doses of diuretics or beta-blockers (usually refers to double max doses) and can not stop dosing
3. atrial fibrillation (AF) or severe arrhythmia
4. severe aortic regurgitation
5. severe thoracic fluids
6. height weight out of ranges: 120-230 cm30-230 kg
7. using more than 3 antihypertensives
8. known secondary hypertension
9. refused to sign informed consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2018-12-31 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline systolic blood pressure at 8 weeks | 8 weeks post-baseline
  Change from baseline systolic blood pressure at 8 weeks in the window of 4-12 weeks
Change from baseline diastolic blood pressure at 8 weeks | 8 weeks post-baseline
  Change from baseline diastolic blood pressure at 8 weeks in the window of 4-12

SECONDARY OUTCOMES:
BP control rate at 8 weeks | 8 weeks post-baseline
  proportion of subjects with BP < 140/90 mmHg at 8 weeks post-baseline visit
Change from baseline heart rate (HR) at 8 weeks | 8 weeks post-baseline
  Change from baseline heart rate (heart beats per minute) at 8 weeks in the window of 4-12 weeks
Change from baseline cardiac index (CI) at 8 weeks | 8 weeks post-baseline
  Change from baseline cardiac index (cardiac output devided by body surface area) at 8 weeks in the window of 4-12 weeks
Change from baseline arterial stiffness (AS) at 8 weeks | 8 weeks post-baseline
  Change from baseline arterial stiffness at 8 weeks in the window of 4-12 weeks
Change from baseline systemic vascular resistance index (SVRI) at 8 weeks | 8 weeks post-baseline
  Change from baseline systemic vascular resistance index at 8 weeks in the window of 4-12 weeks
Change from baseline thoracic blood volume standing/supine ratio (TBR) at 8 weeks | 8 weeks post-baseline
  Change from baseline thoracic blood volume standing vs supine ratio at 8 weeks in the window of 4-12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ningling Sun, Principal Investigator — Department of Hypertension at Heart Centr, Peking University People's Hospital, Beijing, China
Locations (1):
- Peking University People's Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lu Y, Wang L, Wang H, Gu J, Ma ZJ, Lian Z, Zhang Z, Krumholz H, Sun N. Effectiveness of an impedance cardiography guided treatment strategy to improve blood pressure control in a real-world setting: results from a pragmatic clinical trial. Open Heart. 2021 Sep;8(2):e001719. doi: 10.1136/openhrt-2021-001719. PMID 34580169